CLINICAL TRIAL: NCT05141448
Title: Visual Performance of Soft Contact Lenses With Myopia Control Optics
Status: Completed | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CR-6457
Record Dates: First submitted 2021-11-19; First posted 2021-12-02 (Actual); Results first posted 2025-04-08 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Visual Acuity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | Unapproved Device: Yes

ARMS (6):
- Test1/Test2/Control (Experimental): Eligible subjects will be fitted with the run-in lens for approximately one week, then randomized to the sequence Test1/Test2/Control.
  Interventions: Device: 1-Day Acuvue Moist; Device: EMO-118; Device: EMO-114; Device: MiSight® 1 day
- Test1/Control/Test2 (Experimental): Eligible subjects will be fitted with the run-in lens for approximately one week, then randomized to the sequence Test1/Control/Test2.
  Interventions: Device: 1-Day Acuvue Moist; Device: EMO-118; Device: EMO-114; Device: MiSight® 1 day
- Test2/Test1/Control (Experimental): Eligible subjects will be fitted with the run-in lens for approximately one week, then randomized to the sequence Test2/Test1/Control.
  Interventions: Device: 1-Day Acuvue Moist; Device: EMO-118; Device: EMO-114; Device: MiSight® 1 day
- Test2/Control /Test1 (Experimental): Eligible subjects will be fitted with the run-in lens for approximately one week, then randomized to the sequence Test2/Control /Test1.
  Interventions: Device: 1-Day Acuvue Moist; Device: EMO-118; Device: EMO-114; Device: MiSight® 1 day
- Control/Test1/Test2 (Experimental): Eligible subjects will be fitted with the run-in lens for approximately one week, then randomized to the sequence Control/Test1/Test2.
  Interventions: Device: 1-Day Acuvue Moist; Device: EMO-118; Device: EMO-114; Device: MiSight® 1 day
- Control/Test2/Test1 (Experimental): Eligible subjects will be fitted with the run-in lens for approximately one week, then randomized to the sequence Control/Test2/Test1.
  Interventions: Device: 1-Day Acuvue Moist; Device: EMO-118; Device: EMO-114; Device: MiSight® 1 day

INTERVENTIONS:
Device: 1-Day Acuvue Moist — Run-in Contact Lens
Device: EMO-118 — Test Lens1
Device: EMO-114 — Test Lens2
Device: MiSight® 1 day — Control Lens

SUMMARY:
This is a multi-site, bilateral, dispensing, randomized, controlled, single-masked, 3x3 crossover study with a run-in period.

ELIGIBILITY:
Inclusion Criteria:

* Potential subjects must satisfy all of the following criteria to be enrolled in the study:

  1. Read (or be read to) and sign the CHILDREN'S ASSENT (Information and Assent Form) and receive a fully executed copy of the form.
  2. Have parents or legal guardians who must read, understand, and sign the STATEMENT OF INFORMED CONSENT (Parental Permission Form and Authorization to Use and Disclose Medical Information).
  3. Appear able and willing to adhere to the instructions set forth in this clinical protocol.
  4. Be between 7 and 17 (inclusive) years of age at the time of screening.
  5. By self-report, habitually wear soft contact lenses or be a current non-contact lens wearer interested in soft lens wear.
  6. The non-vertex corrected best sphere distance refraction must be between -1.00 D and -4.50 D (inclusive) in each eye.
  7. The magnitude of the cylindrical component of the subject's vertex-corrected distance refraction must be less than or equal to 0.75 D (inclusive) in each eye with any degree of axis.
  8. The distance visual acuity with best sphere distance correction must be 20/25 or better in each eye.
  9. Have ≤ 1.50 D difference in subjective best-sphere refraction between the two eyes.
  10. Have 20/40 or better vision in each eye with wearable spectacles or uncorrected.

      Exclusion Criteria:
* Potential subjects who meet any of the following criteria will be excluded from participating in the study:

  1. Be currently pregnant or lactating.
  2. Be diabetic.
  3. Be currently using any ocular medications. Lubricants (artificial tears) eyedrops are allowed.
  4. Have any current ocular infection of any type.
  5. Have any systemic disease (e.g., Sjogren's Syndrome), allergies, infectious disease (e.g., hepatitis, tuberculosis), contagious immunosuppressive diseases (e.g., HIV), autoimmune disease (e.g., rheumatoid arthritis), any underlying medical condition that makes subjects at risk of severe COVID complications, a history of serious mental illness or seizures, or other diseases, by parent or legal guardian's self-report, which are known to interfere with contact lens wear and/or participation in the study.
  6. Use of systemic medication (e.g., chronic steroid use) that are known to interfere with contact lens wear and/or participation in the study. See section 9.1 for additional details regarding excluded systemic medications.
  7. Have habitually worn rigid gas permeable (RGP) lenses, orthokeratology lenses, or hybrid lenses (e.g. SynergEyes, SoftPerm) within the past 30 days.
  8. Be currently wearing lenses in an extended wear modality.
  9. Be currently wearing soft contact lenses for astigmatism in either eye.
  10. Have participated in a contact lens or lens care product clinical trial within 7 days prior to study enrollment.
  11. Be an employee (e.g., Investigator, Coordinator, Technician) or immediate family member of an employee (including partner, child, parent, grandparent, grandchild or sibling of the employee or their spouse) of the clinical site.
  12. Children who are wards of the State or any other agency, institution, or entity.
  13. Have any ocular allergies, infections, or other ocular abnormalities that are known to interfere with contact lens wear and/or participation in the study. This may include, but is not limited to, entropion, ectropion, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, moderate or above corneal distortion, herpetic keratitis.
  14. Have grade 3 or greater palpebral conjunctival observations or any other grade 2 slit lamp findings on the ISO 11980 classification scale.
  15. Have strabismus (intermittent or constant) or amblyopia.
  16. Have a history or signs of a contact lens-related corneal inflammatory event (e.g., past peripheral ulcer or round peripheral scar).
  17. Have any central corneal scar.
  18. Have a pupil diameter under bright illumination of less than 2 mm in either eye.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 79 (Actual)
Dates: Start 2021-11-22 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Vision Optique, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 79 subjects were enrolled in this study. Of those enrolled, 75 subjects were randomized and dispensed at least one study lens, while 4 subjects failed to meet all eligibility criteria. Of those dispensed, 65 subjects completed the study while, 10 subjects were discontinued from the study.
Groups:
- Run-in Lens/Test 2/Test 1/Control: All subjects wore the Run-in lens during Period 1. Subjects randomized to this arm wore senofilcon A C3 (EMO-114) [Test 2] during Period 2, senofilcon A C3 (EMO-118) [Test 1] during Period 3 and omafilcon A [Control] during Period 4.
- Run-in Lens/Test 2/Control/Test 1: All subjects wore the Run-in lens during Period 1. Subjects randomized to this arm wore senofilcon A C3 (EMO-114) [Test 2] during Period 2, omafilcon A [Control] during Period 3 and senofilcon A C3 (EMO-118) [Test 1] during Period 4.
- Run-in Lens/Test 1/Test 2/Control: All subjects wore the Run-in lens during Period 1. Subjects randomized to this arm wore senofilcon A C3 (EMO-118) [Test 1] during Period 2, senofilcon A C3 (EMO-114) [Test 2] during Period 3 and omafilcon A [Control] during Period 4.
- Run-in Lens/Test 1/Control/Test 2: All subjects wore the Run-in lens during Period 1. Subjects randomized to this arm wore senofilcon A C3 (EMO-118) [Test 1] during Period 2, omafilcon A [Control] during Period 3 and senofilcon A C3 (EMO-114) [Test 2] during Period 4.
- Run-in Lens/Control/Test 2/Test 1: All subjects wore the Run-in lens during Period 1. Subjects randomized to this arm wore omafilcon A [Control] during Period 2, senofilcon A C3 (EMO-114) [Test 2] during Period 3 and senofilcon A C3 (EMO-118) [Test 1] during Period 4.
- Run-in Lens/Control/Test1/Test2: All subjects wore the Run-in lens during Period 1. Subjects randomized to this arm wore omafilcon A [Control] during Period 2, senofilcon A C3 (EMO-118) [Test 1] during Period 3 and senofilcon A C3 (EMO-114) [Test 2] during Period 4.
Period: Period 1
Arm/Group | Run-in Lens/Test 2/Test 1/Control | Run-in Lens/Test 2/Control/Test 1 | Run-in Lens/Test 1/Test 2/Control | Run-in Lens/Test 1/Control/Test 2 | Run-in Lens/Control/Test 2/Test 1 | Run-in Lens/Control/Test1/Test2
Started | 13 | 13 | 15 | 12 | 11 | 11
Completed | 13 | 12 | 15 | 12 | 10 | 11
Not Completed | 0 | 1 | 0 | 0 | 1 | 0
Not completed — Unsatisfactory Visual Response due to Test Article | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Subject No Longer Meets Eligibility Criteria | 0 | 0 | 0 | 0 | 1 | 0
Period: Period 2
Arm/Group | Run-in Lens/Test 2/Test 1/Control | Run-in Lens/Test 2/Control/Test 1 | Run-in Lens/Test 1/Test 2/Control | Run-in Lens/Test 1/Control/Test 2 | Run-in Lens/Control/Test 2/Test 1 | Run-in Lens/Control/Test1/Test2
Started | 13 | 12 | 15 | 12 | 10 | 11
Completed | 13 | 11 | 15 | 11 | 10 | 9
Not Completed | 0 | 1 | 0 | 1 | 0 | 2
Not completed — Unsatisfactory Visual Response due to Test Article | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Subject Withdrawn by PI due to Non Compliance to Protocol | 0 | 0 | 0 | 0 | 0 | 1
Not completed — COVID-19 Related | 0 | 0 | 0 | 1 | 0 | 1
Period: 3
Arm/Group | Run-in Lens/Test 2/Test 1/Control | Run-in Lens/Test 2/Control/Test 1 | Run-in Lens/Test 1/Test 2/Control | Run-in Lens/Test 1/Control/Test 2 | Run-in Lens/Control/Test 2/Test 1 | Run-in Lens/Control/Test1/Test2
Started | 13 | 11 | 15 | 11 | 10 | 9
Completed | 11 | 11 | 15 | 11 | 10 | 8
Not Completed | 2 | 0 | 0 | 0 | 0 | 1
Not completed — Covid-19 related | 2 | 0 | 0 | 0 | 0 | 1
Period: 4
Arm/Group | Run-in Lens/Test 2/Test 1/Control | Run-in Lens/Test 2/Control/Test 1 | Run-in Lens/Test 1/Test 2/Control | Run-in Lens/Test 1/Control/Test 2 | Run-in Lens/Control/Test 2/Test 1 | Run-in Lens/Control/Test1/Test2
Started | 11 | 11 | 15 | 11 | 10 | 8
Completed | 10 | 11 | 15 | 11 | 10 | 8
Not Completed | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Unsatisfactory Visual Response due to Test Article | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All subjects dispensed a study lens.
Groups:
- Total: All subjects dispensed a study lens.
Arm/Group | Total
Number analyzed (Participants) | 75
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: All subjects dispensed a study lens.
  Years | 12.6 (2.36)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: All subjects dispensed a study lens.
  Participants
    Female | 50
    Male | 25
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: All subjects dispensed a study lens.
  Participants
    American Indian or Alaska Native | 0
    Asian | 6
    Native Hawaiian or Other Pacific Islander | 1
    Black or African American | 3
    White | 60
    More than one race | 5
    Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants] — Population: All subjects dispensed a study lens.
  Participants
    United States | 75

OUTCOME MEASURES:

1. Primary Outcome: Binocular Visual Performance (LogMAR)
Description: Visual performance was calculated as binocular contact lens-corrected distance visual acuity using a Logarithm of Minimal Angle of Resolution (logMAR) visual acuity scale. This was evaluated under high luminance and high contrast conditions (HLHC) at 4 meters from Early Treatment Diabetic Retinopathy Study (ETDRS) charts at the 2-week follow-up visit. Lower visual performance values indicate better vision. A value of 0.0 logMAR is equivalent to 20/20 Snellen Visual Acuity. The average visual performance was reported for each lens type. Binocular visual performance for Run-in lens was measured at 1-week follow-up visit.
Time Frame: Up to 2-Week Follow-up
Population: All subjects who successfully completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: logMAR
Groups:
- Run-in: Etafilcon A: Run-in: etafilcon A (1-Week Follow-up)
- Senofilcon A C3 (EMO-114) [Test 2]: Subjects that wore senofilcon A C3 (EMO-114) [Test 2] during any point of the study.
- Senofilcon A C3 (EMO-118) [Test 1]: Subjects that wore senofilcon A C3 (EMO-118) [Test 1] during any point of the study.
- Omafilcon A (MS1D) [Control]: Subjects that wore omafilcon A [Control] during any point of the study.
Arm/Group | Run-in: Etafilcon A | Senofilcon A C3 (EMO-114) [Test 2] | Senofilcon A C3 (EMO-118) [Test 1] | Omafilcon A (MS1D) [Control]
Number analyzed (Participants) | 49 | 49 | 49 | 49
logMAR | -0.10 (0.057) | -0.10 (0.063) | -0.07 (0.064) | -0.11 (0.059)
Statistical Analysis 1: Comparison: Senofilcon A C3 (EMO-118) [Test 1] vs Omafilcon A (MS1D) [Control]; Test type: Non-Inferiority — Non-inferiority was declared if the upper limit of the 95% confidence interval of was below 0.05 logMAR; Linear Mixed Model; Kenward and Roger method was used for denominator degrees of freedom; Mean Difference (Final Values) = 0.04, 95% CI 2-sided [0.02 to 0.06], Standard Error of Mean 0.011 — Mean difference was calculated as senofilcon A C3 (EMO-118) minus omafilcon A

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study. Approximately 2 months per subject.
Description: All subjects dispensed a study lens.
Groups:
- Run-in: Etafilcon A: Subjects that wore the run-in lens, etafilcon A during period 1 of the study.
- Senofilcon A C3 (EMO-114): Subjects that wore senofilcon A C3 (EMO-114) during any point of the study.
- Senofilcon A C3 (EMO-118): Subjects that wore senofilcon A C3 (EMO-118) during any point of the study.
- Omafilcon A: Subjects that wore omafilcon A during any point of the study.
Arm/Group | Run-in: Etafilcon A | Senofilcon A C3 (EMO-114) | Senofilcon A C3 (EMO-118) | Omafilcon A
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/69 | 0/70 | 0/69
Serious Adverse Events (participants affected / at risk) | 0/75 | 0/69 | 0/70 | 0/69
Other Adverse Events (participants affected / at risk) | 0/75 | 0/69 | 0/70 | 0/69

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-29): https://cdn.clinicaltrials.gov/large-docs/48/NCT05141448/Prot_SAP_000.pdf